CLINICAL TRIAL: NCT01643083
Title: Use of Rifaximin in Patients With Functional Dyspepsia: A Randomized Controlled Trial
Brief Title: Rifaximin for Functional Dyspepsia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Wai Keung, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKU_RD1
Record Dates: First submitted 2012-07-15; First posted 2012-07-17 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Functional Dyspepsia
Keywords: Post-prandial distress syndrome
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Active Comparator)
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 400mg tid for 2 wk
  Other Names: Normix
  Arms: Rifaximin
Drug: Placebo — Placebo for 2 week
  Arms: Placebo

SUMMARY:
Functional dyspepsia is a very common medical condition, which occurs in up to 30% of people in the community. However, results of current pharmacological treatment on functional dyspepsia are unsatisfactory. Rifaximin is a minimally absorbed antibiotic that has been used in treatment of non-constipated irritable bowel syndrome (IBS). In particular, bloating and abdominal pain was improved by rifaximin treatment in this group of IBS patients. Whilst there is considerable overlap in symptoms of functional dyspepsia and IBS, the investigators test whether rifaximin is also effective in curing post-prandial distress symptoms related to dyspepsia.

DETAILED DESCRIPTION:
The aim of this study is to test the effects of rifaximin, a minimally absorbed antibiotics, on symptoms of patients with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Non-ulcer dyspeptic patients who fulfill post-prandial distress syndrome according to the Rome III Criteria
* Active dyspeptic symptom
* Normal upper endoscopy
* Urea Breath Test -ve or Rapid urease test -ve
* Not typical gastroesophageal reflux or biliary colic symptoms, but presence of infrequent acid reflux is allowed

Exclusion Criteria:

* No active dyspeptic symptom
* Allergic to rifaximin
* Recent antibiotics use in the past 8 wk
* Recent PPI or H2RA in past 4 wk
* On anti-coagulants, anti-convulsant or oral contraceptives
* On NSAIDs, aspirin or Clopidogrel
* Pregnancy or breast feeding
* Previous gastric surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Adequate relief of dyspeptic symptoms at end of treatment | end of treatment (week 2)
  global symptom improvement

SECONDARY OUTCOMES:
Individual dyspeptic symptom scores | week 2, 4 and 8
  Hong Kong Dyspeptic Index

CONTACTS AND LOCATIONS:
Overall Officials: Wai Keung Leung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

REFERENCES:
- [Derived] Tan VP, Liu KS, Lam FY, Hung IF, Yuen MF, Leung WK. Randomised clinical trial: rifaximin versus placebo for the treatment of functional dyspepsia. Aliment Pharmacol Ther. 2017 Mar;45(6):767-776. doi: 10.1111/apt.13945. Epub 2017 Jan 23. PMID 28112426